CLINICAL TRIAL: NCT03540303
Title: Phase Ⅰ Study of CAR19 T Cells Carrying Cytoplasmic Activated PD-1 in the Treatment of Refractory/Relapsed B Cell Lymphoma
Brief Title: Cytoplasmic Activated PD-1 CAR T Cells in Refractory/Relapsed B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Pregene (ShenZhen) Biotechnology Company, Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH CAR 2-1
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-04

CONDITIONS: Relapsed Non Hodgkin Lymphoma
Keywords: relapsed/refractory, B cell, lymphoma, CAR
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Lymphoma

STUDY DESIGN:
Intervention Model Description: CAR19 T cell therapy improves the clinical efficacy of refractory/relapsed B-cell lymphoma, and the combined PDL1 inhibitors may further improve the efficacy of CD19 CART in the treatment of lymphomas. The clinical efficacy of KITE's CAR19 T cells and PD-L1 inhibition was reported. This phase 1 study was conducted in 9 patients with DLBCL, 8 patients got remission and during which 5 got complete remission. However, this type of treatment requires more data and observation in a larger sample of patients. In addition, Kite Pharmaceuticals' CD19 CART is priced at 370,000 US dollars. The cost of immune checkpoint inhibitors is also very expensive. Only very small proportion of patients could afford for that expenses. In this study, genetically engineered CAR T cells, which carry cytoplasmic activated PD1, are not inhibited by PDL1 molecules, will avoid the simultaneous application of immune checkpoint antibodies and the according adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR19 T cells carrying cytoplasmic activated PD-1 (Experimental): patients with refractory/relapsed B-NHL receive a preconditioning before infusion of CAR T cells.
  Interventions: Drug: CAR19 T cells carrying cytoplasmic activated PD-1

INTERVENTIONS:
Drug: CAR19 T cells carrying cytoplasmic activated PD-1 — step 1: Collect 50-100ml of peripheral blood for culture of CAR19 T cells carrying cytoplasmic activated PD-1 step 2. After 72 hours, pretreated with FC regimen, details as follow Cyclophosphamide 600-800mg/m2 for 2 days Fludarabine 25-30mg/m2 for 3 days step 3: After another 48 hours transfusion the cells back to the patients the numbers of infused CAR T cells are 2x106 /kg for the first 3 patients, 6x106 /kg for the second 3 patients and 18x106 /kg for the third 3 patients.
  After finishing this, another 6 patients will be enrolled for observation of efficacy.

SUMMARY:
Evaluation of the safety and efficacy of CAR19 T cells carrying cytoplasmic activated PD1 in patients with refractory relapsed B-cell lymphoma

DETAILED DESCRIPTION:
Although CAR19 T cell therapy brings hope, the patients with refractory/relapsed B-cell lymphoma is still a problem for the current treatment. There are still some patients with poor therapeutic efficacy, and the efficacy of CAR19-T cell therapy remains to be improved. Basic research shows that there is a synergistic effect between CAR-T cell therapy and anti-PD1 pathway, and it did have efficacy in clinic. However, the regimen of CAR19-T cells combined anti-PD1 inhibitors need to be combined with the application of anti-PD1 antibody and culture of CART cells during the treatment, there may be adverse events to PD1 antibodies. In this study, CAR19T cells carrying cytosolic activated PD1 possess the dual effects of CAR19T cells and anti-PD1 or anti-PD-L1 antibodies while overcoming the adverse events of anti-PD1 inhibitors, and might have better efficacy than conventional CAR19T cells plus anti-PD1 or anti-PD-L1 antibody treatment, with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old and the expected lifetime >3 months
* Refractory/relapsed CD19 positive B cell lymphoma by pathology
* ECOG score <2
* Measureable lesions according to RECIST 1.1
* Sufficient heart, liver, kidney and bone marrow function (heart: no heart disease or coronary heart disease, patient heart function NYHA grade 1-2; liver: TBIL ≤ 3ULN, AST ≤ 2.5ULN, ALT ≤ 2.5ULN; kidney: Cr≤ 1.25ULN; bone marrow: WBC ≥ 2.0 × 109/L, Hb ≥ 80 g/L, PLT ≥ 30 × 109/L)
* no serious allergies
* No other serious diseases that conflict with this protocol (eg, autoimmune diseases, immunodeficiency, organ transplantation)
* No other history of malignancy
* No serious mental disorders
* Women of childbearing age must be negative for blood pregnancy test within 7 days and must take appropriated contraceptive measures during and 3 months after the study
* The patient himself agrees to participate in this clinical study and signed the "informed consent"

Exclusion Criteria:

* Lactating women
* Severe infectious or viral diseases (HIV positive, syphilis, etc.)
* Active hepatitis B or C viral hepatitis
* Patients who used high-dose glucocorticoids within 1 week
* Participation in other clinical studies in the past 3 months or having been treated with other gene products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
safety: occurrence of study related adverse events | 6 months
  occurrence of study related adverse events

SECONDARY OUTCOMES:
objective response rate | 3 months and 6 months
  tumor burdens shrink more than 30 percent by RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, M.D, Study Chair — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China